CLINICAL TRIAL: NCT04559490
Title: Formula - Understanding Nutrition (FUN)
Brief Title: Baby Formula and Health
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Bridget Young, Assistant Professor, University of Rochester
Other Study IDs: STUDY00004724
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Pancreas Disease
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard formula: Participants receiving intact protein lactose-based formula, exclusively for at least 3 months.
- Sensitive: Participants receiving intact protein glucose/sucrose- based formula, exclusively for at least 3 months.

SUMMARY:
The purpose of this study is to learn about how different types of carbohydrates used in infant formula may affect a baby's intestines and pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Mothers ≥ 19 years of age
* Singleton birth
* Healthy Infants
* Infant between 3-6 months at the time of visit and exclusively fed one of the formulas for a minimum of 3 months

Exclusion Criteria:

* Delivery before 35 weeks
* Infant birth weight <2500g
* Infants exhibiting growth faltering (loss of more than 25 percentile points) between 1 month to the time of study visit for either weight or length.
* Infant medical or genetic indications that would impact normal feeding behavior, insulin signaling or growth patterns.
* Infant consumption of more than two servings of complementary foods per day before the study visit.

Min Age: 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mothers and infants will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2023-09-16 (Actual)

PRIMARY OUTCOMES:
mean change in blood glucose | baseline to 1 hour
  change in blood glucose from fasting to 1 hour post glucose challenge

SECONDARY OUTCOMES:
mean endogenous insulin secretion | baseline to 1 hour
  change in mean insulin collected at baseline and 1 hour post glucose challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center of the University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided